CLINICAL TRIAL: NCT01761474
Title: Carbon Dioxide Insufflations vs. Air Insufflation in Therapeutic ERCP: A Randomized Double-blind Comparative Study Depending on Sedation Methods
Brief Title: CO2 Versus O2 Insufflation During ERCP Depending on Sedation Protocols
Status: Completed | Type: Observational
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae Hoon Lee, Professor, Soon Chun Hyang University
Other Study IDs: ERCP-Sedation
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Satisfaction; Complication
Keywords: Carbon dioxide insufflation; Air insufflatioin; ERCP; Sedation
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1. Carbon dioxide insufflation with BPS: Both midazolam (0.05 mg/kg body weight; 1 mg if age[70 or ASA class III-IV) and fentanyl (50 lg; 25 lg if age[70 or ASA class III-IV) were given intravenously at the initiation of sedation. Thereafter, repeated doses of 10-20 mg propofol were administered to achieve a moderate level of sedation. Maintenance of sedation was also performed with repeated doses of 10-20 mg propofol.
- 2. Carbon dioxide insufflation with Propofol: Sedation was induced by intravenous bolus injection of propofol (0.5 mg/kg body weight; 10 mg if age[70 or ASA class III-IV), followed by repeated doses of 10-20 mg propofol to induce sedation. Repeated doses of 10-20 mg propofol were then administered to maintain adequate sedation, according to the desired sedation depth and patient risk profile.
- 3. Air insufflation with BPS: Both midazolam (0.05 mg/kg body weight; 1 mg if age[70 or ASA class III-IV) and fentanyl (50 lg; 25 lg if age[70 or ASA class III-IV) were given intravenously at the initiation of sedation. Thereafter, repeated doses of 10-20 mg propofol were administered to achieve a moderate level of sedation. Maintenance of sedation was also performed with repeated doses of 10-20 mg propofol.
- 4. Air insufflation with Propofol: Sedation was induced by intravenous bolus injection of propofol (0.5 mg/kg body weight; 10 mg if age[70 or ASA class III-IV), followed by repeated doses of 10-20 mg propofol to induce sedation. Repeated doses of 10-20 mg propofol were then administered to maintain adequate sedation, according to the desired sedation depth and patient risk profile.

SUMMARY:
Endoscopic retrograde cholangiopancreatography(ERCP) and related procedures can cause abdominal pain and discomfort. Some clinical trials have indicated, using the visual analogue scale (VAS) score, that CO2 insufflation during ERCP ameliorates the suffering of patients without complications, compared with air insufflation. However, differences in patient suffering between CO2 and air insufflation after ERCP depending on sedation protocols have not been reported. We therefore planned prospective, double-blind, randomized, controlled study with CO2 and air insufflation during ERCP depending on sedation protocol.

ELIGIBILITY:
Inclusion Criteria:

* candidates for therapeutic ERCP

Exclusion Criteria:

* age<18 years
* pregnant women
* total gastrectomy
* uncontrolled coagulopathy
* American Society of Anesthesiologist(ASA) Class V
* neurologic impairment
* known allergy to the drugs used
* history of complications with previous sedation, sedative
* alcohol abuse
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study had an 80% power to detect a 20% difference in PAIN score any two groups, assuming 2-sided tests at a 5% significance level.Assuming a 10 % dropout rate, 220 patients were needed.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sedation quality | After patients' alertness (at least 10 minutes later), 3 hrs, and 24 hrs later
  Abdominal pain, discomfort, and gas accumulation

SECONDARY OUTCOMES:
Complications | After completion of procedures (within 2 hrs) and 24 hrs later
  Procedure related complications; pancreatitis, bleeding, cholangitis, or perforation
Procedure outcome | After completion of procedure, within 2hrs
  1. Technical success or fail of procedure
  2. Procedure quality and satisfaction to patients and endoscopist

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hoon Lee, PhD, Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Soon Chun Hyang University Cheonan Hospital, Cheonan, Chungchungnam-do, South Korea